CLINICAL TRIAL: NCT01559025
Title: Evaluation of Vildagliptin (Galvus®) as add-on to Insulin in Residual β-cell Function and Inflammatory Markers in New-onset Type 1 Diabetes Mellitus.
Brief Title: Evaluation of Vildagliptin (Galvus®) as add-on to Insulin in New-onset Type 1 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Tatiana Valente, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ABR01T
Record Dates: First submitted 2011-11-30; First posted 2012-03-20 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes; Insulin Dependent Diabetes; Juvenile Onset Diabetes Mellitus; Autoimmune Diabetes
Keywords: Type 1 diabetes; Vildagliptin; Galvus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Vildagliptin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin therapy (No Intervention): Patients will receive the conventional treatment with insulin
- Vildagliptin (Active Comparator): Patients will receive vildagliptin besides the conventional treatment with insulin
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin ( Galvus 50mg twice day) during one year
  Other Names: Galvus; DPP-4 inhibitor
  Arms: Vildagliptin

SUMMARY:
The primary objective of this study is to evaluate the action of DPP-IV inhibitors in the prevention of progressive beta cell dysfunction in patients with type 1 diabetes mellitus newly diagnosis ( less than 6 months).

The secondary objectives are:

1. To define the immune and inflammatory profile
2. To define the secretion of glucagon and GLP-1
3. To assess the glycemic variability

DETAILED DESCRIPTION:
Clinical and autopsy studies show that up to 30% of patients with type 1 diabetes mellitus show a detectable β-cell function at clinical diabetes. The preservation of this endogenous insulin production, even if it is small, can have a great impact on the evolution of long-term disease through improving glycemic control, reducing chronic diabetes complications and hypoglycemia. Strategies for preventing the loss of beta cell are based on stopping the autoimmune process and also in the preservation and regeneration of beta cells. Currently have been questioned the potential use of GLP-1 for new-onset type 1 diabetes. The justification for this issue is based on the fact that this class of drugs, besides acting on insulin secretion and glucose regulation, may be effective to preserve and expand beta cell mass, which has been shown in animals. Ideal candidates for this treatment are newly diagnosed patients who still have significant viable beta cell mass.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 35 years
* Up to 6 months of clinical diagnosis
* Fasting C-peptide ≥ 0.25 ng / ml
* HbA1C <9.0%
* Positive autoantibodies (anti-GAD, Anti-Insulin and Anti-IA2)
* Without chronic complications

Exclusion Criteria:

* Hepatic, cardiac, pulmonary and hematologic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Beta cell function | C peptide will be measured by the area under the curve of stimulated C peptide within the first 2 hours every 3 months up to one year
  The primary objective of this study is to evaluate the action of DPP-IV inhibitors in the prevention of progressive beta cell dysfunction in patients with type 1 diabetes mellitus newly diagnosis ( less than 6 months). It will be measured by the area under the curve of stimulated C peptide within the first 2 hours

SECONDARY OUTCOMES:
Immune and inflammatory profile | 0,3,6,9,12th months
  Inflammatory profile will be measured by some markers such as TNF-alpha, IL-10 and PCR.
  Immune profile will be obtained by the expression of FOXP3 in both groups.
Secretion of Glucagon and GLP-1 | 0,3,6, 9 and 12months
  It will be obtained by the measure of glucagon and GLP-1 levels
Glycemic variability | 0, 6 and 12months
  To evaluate the glycemic variability, it will be installed the continuos glucose monitoring system (CGMS) for seven days during the 0, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Dib, Principal Investigator — FUSãoPaulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil